CLINICAL TRIAL: NCT03715582
Title: PROSPECTIVE ANALYSIS BETWEEN TRIMETAZIDINE Versus PLACEBO IN MYOCARDIAL INJURY AFTER PERCUTANEOUS CORONARY INTERVENTION IN PATIENTS WITH INSTANT ANGINA AND DIABETES MELLITUS
Brief Title: Trimetazidine in Myocardial Injury After Percutaneous Coronary Intervention in Patients With Angina and Diabetes
Acronym: Trimeta
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSInCor-Trimetazidine
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus; Angina, Unstable
MeSH Terms: conditions — Diabetes Mellitus; Angina, Unstable | interventions — Trimetazidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trimetazidine (Experimental): The randomization will be done with a list generated by the central pharmacy of the Hospital das Clínicas, Medical School, USP. When the patient is randomized to the trimetazidine pill group, he / she will initiate the medication at 70 mg oral dose (2 tablets of Vastarel ® MR 35 mg single dose) 2 hours before the procedure.
  Interventions: Drug: trimetazidine
- placebo (Experimental): The randomization will be done with a list generated by the central pharmacy of the Hospital das Clínicas, Medical School, USP. When randomized to the placebo oral tablets group, the patient will receive placebo (orally, 2 single dose tablets) also 2 hours prior to PCI.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: trimetazidine — Pills of masking drug - trimetazidine
  Arms: trimetazidine
Drug: Placebo Oral Tablet — Pills of masking drug - placebo
  Other Names: placebo
  Arms: placebo

SUMMARY:
Introduction: Recent studies have suggested that trimetazidine may help reduce myocardial damage following percutaneous coronary intervention. However, the evaluation of the potential of this medication in the reduction of myocardial damage in patients with diabetes mellitus and unstable angina, in a prospective and randomized way, has not yet been described. Objective: The aim of this study was to evaluate the efficacy and safety of the use of trimetazidine versus placebo in patients with diabetes mellitus and unstable angina undergoing coronary stent angioplasty. Methodology: For this, a unicentric, randomized, double blind and prospective study will be performed in a comparative manner. Hospital data (test results, medical outcomes, drug dose, complications) of patients will be analyzed for safety and effectiveness. Myocardial damage will be measured by means of ultrasensitive Troponin dosages. Expected results: The use of trimetazidine reduces myocardial damage in patients with diabetes mellitus and unstable angina undergoing coronary stent angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women aged> 18 years.
* Diagnosis of unstable angina with chest pain at least 2 hours after arrival at the emergency unit.
* Measurement of troponin less than the upper limit of the normality of the method.
* Indication of cardiac catheterization and need for percutaneous coronary intervention with uniarterial stent within 24 hours of admission.
* No known allergy to trimetazidine.
* Prior diagnosis of diabetes mellitus under specific treatment.
* ClCr> 30 mL / min.
* Signed consent form.

Exclusion Criteria:

* Pregnancy.
* Hemodynamic instability (pulmonary congestion / systolic blood pressure less than 90 mmHg).
* SCA with ST elevation or troponin elevation.
* Body mass index greater than 40 kg / m2.
* Use of oral anticoagulant.
* Orotracheal intubation.
* Left ventricular outflow tract obstruction.
* Allergy to iodinated contrast.
* Thoracic trauma in the last 30 days.
* Previous surgical myocardial revascularization.
* Presence of ventricular arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
peak values of troponin and CKMB after PCI | 24 hours
  comparing groups for peak values of troponin and CKMB after PCI.

SECONDARY OUTCOMES:
peak values of CRP | 24 hours
  Comparison between groups for peak values of CRP after PCI.
peak values of creatinine | 24 hours
  Comparison between groups for peak values of creatinine after PCI.
peak values of leukogram | 24 hours
  Comparison between groups for peak values of leukogram after PCI.
occurrence of sustained ventricular arrhythmia | 24 hours
  Combined comparison between the occurrence of sustained ventricular arrhythmia
occurrence of cardiogenic shock, | 24 hours
  Combined comparison between the occurrence of cardiogenic shock,
occurrence of cardiorespiratory arrest, | 24 hours
  Combined comparison between the occurrence of cardiorespiratory arrest
occurrence of worsening of renal function | 24 hours
  Combined comparison between the occurrence of worsening of renal function (increase of 0.5 mg / dL in relation to admission creatinine or 25% above baseline)
occurrence of need for reintervention | 24 hours
  Combined comparison between the occurrence of need for reintervention
occurrence of cerebrovascular accident | 24 hours
  Combined comparison between the occurrence of cerebrovascular accident
occurrence of death | 24 hours
  Combined comparison between the occurrence of death

CONTACTS AND LOCATIONS:
Overall Officials: Mucio Tavares, MD, Principal Investigator — Unidade Clínica de Emergência
Locations (1):
- Instituto do Coração - HMFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided